CLINICAL TRIAL: NCT06182657
Title: The Prognostic Value of the Degree of Pathological Response at One Cycle of Induction Chemotherapy for Locally Advanced Nasopharyngeal Carcinon-a Prospective Observational Study
Brief Title: The Prognostic Value of the Degree of Pathological Response of Induction Chemotherapy for NPC
Status: Recruiting | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NPC-pCR
Record Dates: First submitted 2023-07-20; First posted 2023-12-27 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-07

CONDITIONS: Nasopharyngeal Carcinoma; Pathologic Complete Response; Tumor Microenvironment
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the prognostic value of pathological remission after one cycle of induction chemotherapy in locally advanced nasopharyngeal carcinoma, and the change of immune micro-environment after one cycle induction chemotherapy, including the density of immune cells infiltration and tertiary lymphoid structures.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to sign informed consent
2. Age > 18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (amend based on specific study)
4. Histological confirmation of NPC (regardless if EBER positive or negative)
5. Locally advanced NPC, UICC stage III-IVa
6. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
2. Distant metastases
3. Prior systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, radiotherapy, biologic therapy, tumour embolization, monoclonal antibodies) of the locally advanced NPC.
4. History of another primary malignancy
5. Female patients who are pregnant
6. Known allergy or hypersensitivity to any drugs
7. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven stage III-IVA NPC (according to the 8th edition of Union for International Cancer Control stage classification).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  PFS is defined as the time from treatment to date of first documentation of progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  OS is defined as the time from treatment to death, regardless of disease recurrence.
Distant metastasis-free survival (DMFS) | 3 years
  DMFS is defined as the time from diagnosis to the date of distant metastasis or when censored at the latest date.
Pathological complete response (pCR) rate | At the end of Cycle 1 (each cycle is 21 days).
  pCR is defined as the absence of residual invasive.
Infiltrating Immune cell density | At the end of Cycle 1 (each cycle is 21 days).
  CD3+ T cells, CD8+ T cells, CD20+ B cell and Tertiary lymphoid structure

CONTACTS AND LOCATIONS:
Overall Officials: Jingao Li, PhD, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jingao Li, Nanchang, Jiangxi, China